CLINICAL TRIAL: NCT03319719
Title: Evaluation of Pain With Belotero® Balance With Integral Lidocaine for Correction of the Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M930021001
Record Dates: First submitted 2017-10-04; First posted 2017-10-24 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2018-01

CONDITIONS: Correction of Moderate to Severe Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Belotero® Balance with integral lidocaine (Experimental): Belotero® Balance with integral lidocaine will be injected in one of the two NLF (split-face study design: treatment side will be randomized)
  Interventions: Device: Belotero® Balance with integral lidocaine
- Belotero Balance without lidocaine (Active Comparator): Belotero Balance without lidocaine will be injected in one of the two NLF (split-face study design: treatment side will be randomized)
  Interventions: Device: Belotero® Balance

INTERVENTIONS:
Device: Belotero® Balance with integral lidocaine — Mode of application: intradermal injection. Maximum treatment volume: 3 mL per nasolabial fold over two Treatment sessions.
  Other Names: Hyaluronic acid dermal filler with lidocaine, single use syringe
  Arms: Belotero® Balance with integral lidocaine
Device: Belotero® Balance — Mode of application: intradermal injection. Maximum treatment volume: 3 mL per nasolabial fold over two Treatment sessions.
  Other Names: Hyaluronic acid dermal filler, single use syringe
  Arms: Belotero Balance without lidocaine

SUMMARY:
Demonstrate the effectiveness of Belotero Balance with lidocaine (Test group) for the reduction of injection-related pain in comparison to Belotero Balance without lidocaine (Control group) for the correction of NLFs.

Identify and describe adverse events (AEs) and serious adverse events (SAEs) during the course of the study. Additionally, common treatment site responses (CTRs) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Has right and left NLF ratings of 2 or 3 (moderate or severe) on the Merz NLF Scale, as determined by the blinded evaluator.
2. Has the same Merz NLF Scale rating on both NLFs (i.e., symmetrical NLFs).
3. Is at least 18 years of age.
4. Understands and accepts the obligation not to receive any other procedures (i.e., dermal fillers, toxin treatments, facial ablative or fractional laser, microderm abrasion, chemical peels, non-invasive skin-tightening [e.g., Ultherapy, Thermage], or surgical procedures) below the orbital rim on the face during study participation.

Exclusion Criteria:

1. Had prior surgery in the mid- and/or lower-face area, including the nasolabial fold(s), or has a permanent implant or graft in the mid- and/or lower-face area that could interfere with effectiveness assessments. (NOTE: Rhinoplasty is permitted if the procedure was ≥ 12 months prior to study enrollment.)
2. Has skin or fat atrophy, beyond typical for the subject's age, in the mid- to lower-facial region or has been diagnosed with a connective tissue disorder.
3. Has unphysiological skin laxity or sun damage, beyond typical for the subject's age, or subject plans to tan during the study period.
4. Has undergone oral surgery (e.g., orthodontia, extraction, implants) in the past 30 days or plans to receive such surgery during participation in the study.
5. Has received mid- and/or lower-facial region treatments with porcine-based collagen fillers, Belotero® Volume, JUVÉDERM VOLUMA®, Restylane® Lyft, RADIESSE®, poly L-lactic acid (PLLA), or mesotherapy within the past 24 months and/or with other hyaluronic acid (HA) products within the past 12 months or plans to receive such treatment during participation in the study.
6. Has ever been treated with fat injections or permanent and/or semi-permanent dermal fillers in the mid- and/or lower-facial region or plans to receive such treatment during participation in the study.
7. Has received immunosuppressive medications or systemic steroids (except intranasal/inhaled steroids) in the past 2 months or plans to receive such treatment during participation in the study.
8. Has an acute inflammatory process or infection at the injection site (e.g., skin eruptions such as cold sores, cysts, pimples, acne, eczema, hives, streptococcus infections) or history of chronic or recurrent infection or inflammation with the potential to interfere with study results or increase the risk of AEs.
9. Has a history of allergic/anaphylactic reactions, including hypersensitivity to lidocaine or anesthetics of the amide type, hyaluronic acid preparations, gram positive bacterial proteins, or any of the device components.
10. Has a known bleeding disorder or has received or is planning to receive anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti-inflammatory drugs (oral/injectable corticosteroids or NSAIDs [e.g., aspirin, ibuprofen]), or other substances known to increase coagulation time (e.g., vitamins or herbal supplements, i.e., Vitamin E, garlic, gingko) from 10 days before injection to 3 days after injection.
11. Has any other medical condition with the potential to interfere with study outcome assessments or compromise subject safety (i.e., increase the risk of adverse events).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kreymerman, MD, FACS, Study Director — Merz North America, Inc.
Locations (3):
- United States (3):
  - Center for Dermatology and Dermatology Surgery; Merz Investigational Site #0010170, Washington D.C., District of Columbia
  - Tennessee Clinical Research Center; Merz Investigational Site #0010097, Nashville, Tennessee
  - Research Across America (Synexus); Merz Investigational Site #0010125, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 investigative sites in the United States.
Pre-assignment Details: A total of 65 participants were screened, out of which 52 participants were randomized and treated. Of these, 51 participants completed the study.
Groups:
- Belotero Balance With or Without Lidocaine: Participants received treatment with Test Product belotero balance with lidocaine (BBL), injection, in one of the two nasolabial fold (NLF) and Control Product belotero balance (BB) without lidocaine, injection, in the contralateral NLF on Day 1. The BBL and BB injections were given in the alar-targus line to the oral commissure. The maximum treatment volume was 3 milliliter (mL) per NLF over two treatment sessions, on Day 1 and optional touch-up at Week 2. Participants who were eligible for an optional touch-up treatment to achieve optimal correction based on investigator's discretion received the BBL and BB injections on Week 2.
Period: Overall Study
Arm/Group | Belotero Balance With or Without Lidocaine
Started | 52
Completed | 51
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) included all participants who were enrolled into the study, randomized, and received an injection.
Groups:
- Belotero Balance With or Without Lidocaine: Participants received treatment with Test Product BBL, injection, in one of the two NLF and Control Product BB without lidocaine, injection, in the contralateral NLF on Day 1. The BBL and BB injections were given in the alar-targus line to the oral commissure. The maximum treatment volume was 3 mL per NLF over two treatment sessions, on Day 1 and optional touch-up at Week 2. Participants who were eligible for an optional touch-up treatment to achieve optimal correction based on investigator's discretion received the BBL and BB injections on Week 2.
Arm/Group | Belotero Balance With or Without Lidocaine
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic and not Latino | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 16
  Caucasian | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Skin type I = white; very fair, red or blonde hair blue eyes; freckles; always burns, never tans, skin type II = white, fair, red or blond hair; blue, hazel or green eyes; usually burns, tans with difficulty, skin type III = cream white; fair with any eye or hair color (common); sometimes mild burn, gradually tans, skin type IV = brown; typical Mediterranean Caucasian skin; rarely burns, tans with ease, skin type V = dark brown; mid-eastern skin types; very rarely burns, tans easily, and skin type VI = black; never burns, tans very easily.
  Participants
    Skin Type I | 1
    Skin Type II | 20
    Skin Type III | 15
    Skin Type IV | 4
    Skin Type V | 5
    Skin Type VI | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Using Visual Analog Scale (VAS)
Description: Pain was assessed using a using a 10 centimeter (cm) VAS. It included 21-numbered circles at 0.5 cm increments, spanning 10 cm total, and was anchored by word descriptors. The VAS scores ranged from 0 (no pain) to 10 (very severe pain).The level of pain was evaluated for each NLF independently immediately upon completion of injection (time zero) on Day 1.
Time Frame: Day 1
Population: The full analysis set (FAS) included all randomized participants and were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Test Product: BBL: Participants received treatment with Test Product BBL, injection, in one of the two NLF on Day 1. The BBL injections were given in the alar-targus line to the oral commissure. The maximum treatment volume was 3 mL per NLF over two treatment sessions, on Day 1 and optional touch-up at Week 2. Participants who were eligible for an optional touch-up treatment to achieve optimal correction based on investigator's discretion received the BBL injection on Week 2.
- Control Product: BB: Participants received treatment with Control Product BB without lidocaine, injection, in the contralateral NLF on Day 1. The BB injections were given in the alar-targus line to the oral commissure. The maximum treatment volume was 3 mL per NLF over two treatment sessions, on Day 1 and optional touch-up at Week 2. Participants who were eligible for an optional touch-up treatment to achieve optimal correction based on investigator's discretion received the BB injection on Week 2.
Arm/Group | Test Product: BBL | Control Product: BB
Number analyzed (Participants) | 52 | 52
score on a scale | 3.07 (1.88) | 5.94 (2.41)
Statistical Analysis 1: Comparison: Test Product: BBL vs Control Product: BB; Test type: Superiority; p < 0.0001, t-test, 2 sided — p-value from paired two-sided t-tests of no difference between test and control groups; Mean Difference (Net) = -2.88, 95% CI 2-sided [-3.42 to -2.33]

2. Secondary Outcome: Percentage of Responders With Greater Than or Equal to (>=) 1-point Improvement as Evaluated Using Merz NLF Scale at Week 6
Description: The Merz NLF scale was used to measure the aesthetic effectiveness of the study products. Each NLF was assessed separately. The Merz NLF scale is a 5-grade scale ranging from 0 (no folds) to 4 (very severe folds). Response was defined >=1-point improvement on the Merz NLF Scale for each NLF compared to baseline.
Time Frame: Week 6
Population: The FAS included all randomized participants and was analyzed as randomized. Participants who were evaluable for this measure at given time period were included.
Measure: Number; unit: percentage of participants
Arm/Group | Test Product: BBL | Control Product: BB
Number analyzed (Participants) | 51 | 51
percentage of participants | 51.0 | 52.9

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to Week 6
Population: The SES included all participants who were enrolled into the study, randomized, and received an injection.
Measure: Number; unit: participants
Arm/Group | Belotero Balance With or Without Lidocaine
Number analyzed (Participants) | 52
participants
  TEAEs | 5
  SAEs | 0

4. Secondary Outcome: Number of Participants With Incidence of Any Common Treatment Site Response (CTR) Evaluated Using Participant Diaries
Description: CTR were evaluated using participant diaries. Participants recorded daily in the diary any pre-defined CTR that occurred. These CTR included swelling, firmness, lumps/bumps, bruising, pain, tenderness upon pressing, redness, discoloration (not redness or bruising), itching, stinging/burning, and numbness.
Time Frame: Baseline up to Week 6
Population: The SES included all participants who were enrolled into the study, randomized, and received an injection.
Measure: Number; unit: participants
Arm/Group | Test Product: BBL | Control Product: BB
Number analyzed (Participants) | 52 | 52
participants | 41 | 45

5. Secondary Outcome: Number of Participants With Incidence of Any CTR by Severity Evaluated Using Participant Diaries
Description: as for outcome 4
Time Frame: Baseline up to Week 6
Population: The SES included all participants who were enrolled into the study, randomized, and received an injection. Participants who were evaluable for this measure at given time period were included.
Measure: Number; unit: participants
Arm/Group | Test Product: BBL | Control Product: BB
Number analyzed (Participants) | 52 | 52
participants
  Mild | 23 | 24
  Moderate | 14 | 18
  Severe | 4 | 3

6. Secondary Outcome: Number of Participants With Incidence of Any CTR by Duration Evaluated Using Participant Diaries
Description: as for outcome 4
Time Frame: Baseline up to Week 6
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Test Product: BBL | Control Product: BB
Number analyzed (Participants) | 52 | 52
participants
  1 to 3 days | 16 | 20
  4 to 7 days | 14 | 14
  8 to 17 days | 8 | 9
  15 to 30 days | 3 | 2
  Greater than (>) 30 days | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 6
Description: The investigator queried the participant for adverse events at each visit.
Arm/Group | Belotero Balance With or Without Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 5/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belotero Balance With or Without Lidocaine (N=52)
Headache (Nervous system disorders) | 2
Gastroenteritis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT03319719/SAP_000.pdf
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT03319719/Prot_001.pdf